CLINICAL TRIAL: NCT01181843
Title: A Prospective, Observational, Double-blind (Black-Box) Study Evaluating Incidence, Severity and Predictive Factors of Respiratory Depression During Postoperative Neuraxial Opioid Analgesia in Obstetric Patients After Cesarean Delivery Using Current Standard Intermittent Postoperative Monitoring Compared to Continuous Pulse Oximetry / Capnography
Brief Title: Incidence of Respiratory Depression in Cesarean Section
Status: Terminated | Type: Observational
Why Stopped: departmental financial support withdrawn
Sponsor: Wake Forest University (Other)
Collaborators: Forsyth Medical Center (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: FMC IRB 2010.200
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-02

CONDITIONS: Respiratory Depression; Postoperative Pain
Keywords: postoperative pain management; respiratory depression; capnography; duramorph
MeSH Terms: conditions — Respiratory Insufficiency; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cesearean sections receiving duramorph

SUMMARY:
This study is designed to determine the incidence and severity of respiratory depression in elective cesarean section patients who have received a spinal or epidural narcotic called duramorph for management of postoperative pain. A monitoring device called a capnograph as well as a device called a pulse oximeter is placed on the patient once in the recovery room after delivery. The capnograph monitors the carbon dioxide level that the patient breathes out as well as their respiratory rate. The pulse oximeter is a device that is taped on the patient's finger and measures their oxygen saturation level. The monitoring is maintained for 18-24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Are female >= 18 years of age and <=55 years of age with ASA class I-III
* Schedule for cesarean surgery
* Are willing and able to sign informed consent form for this study
* Are willing and able to follow the instruction in this study protocol

Exclusion Criteria:

* Have known contraindication/allergy to neuraxial anesthesia or morphine.
* Have an ASA class > III
* Age > 55 years

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects having an elective cesearean section and having as their anesthetic either a spinal or epidural and receiving duramorph
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
RESPIRATORY DEPRESSION | 24 HOURS
  RESPIRATORY DEPRESSION OBSERVATION ONLY OF CURRENT PRACTICES, DOES NOT INVOLVE TREATMENT

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center-Dept of OB Anesthesia, Winston-Salem, North Carolina, United States